CLINICAL TRIAL: NCT06885983
Title: Cellular and Tissue Mechanisms of Bone and Soft Tissue Healing After Augmentation of Alveolar Ridge With Cross-linked Type I Collagen Membrane
Brief Title: Healing After Augmentation of Alveolar Ridge Using Collagen Membrane
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Bozidar Brkovic, DDS, MSc, PhD, Professor, Full professor, University of Belgrade
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 36/39/24
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Bone Healing; Augmentation; Augmentation, Alveolar Ridge
Keywords: Implantation; Augmenatation; CROSS-LINKED TYPE I COLLAGEN MEMBRANE

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implant placement with augmentation (Experimental): Patients who are indicated for implant rehabilitation. Guided tissue regeneration employs augmentation with cross-linked type I collagen membrane to create different gingiva phenotype. The material will be placed after implantation using the following standard surgical protocols. Collagen membrane will serve as a barrier for epithelial cells and thereby promote bone healing.
  Interventions: Procedure: implant placement; Procedure: Guided bone regeneration
- Implant placement without augmentation (Active Comparator): Patient that needs implant placement in order for functional and aesthetic rehabilitation. Surgical procedures done in this group follow standard surgical protocols for implant placement without regenerative therapy.
  Interventions: Procedure: implant placement

INTERVENTIONS:
Procedure: implant placement — Late implant placement without regenerative therapy
Procedure: Guided bone regeneration — Application of collagen membrane after implant placement.
  Arms: Implant placement with augmentation

SUMMARY:
One of the prerequisites for successful prosthetic implant therapy of patients is achieving the initial stability of the embedded implant, which largely depends on the width alveolar ridge, at the place of its installation. Regenerative therapy of the horizontal dimension of the alveolar ridge simultaneously with the installation of implants is carried out using biocompatible materials; a basket of thin ones substitutes and collagen membranes. Clinical application of the collagen matrix to date has shown successful regeneration soft tissue in corrective surgery of the oral mucosa, by increasing the volume of the gingiva, approximately as effective as the application of a connective tissue graft from the palate. In the current literature, there is no data on the cellular effects of the regeneration of soft, a especially bone tissue, after the application of a membrane with cross-linked collagen type I, u regenerative therapy of fenestrations, dehiscence and buccal contour augmentations bone lamellae, simultaneously with implant placement. Also, tissue monitoring mechanisms of regeneration of soft and bone tissue, has not been shown in the literature so far controlled and systematized results using the Primescan digital program scans and software analysis of soft tissue regeneration parameters, as well as their own correlations with CBCT and clinical analysis.

DETAILED DESCRIPTION:
The physiological process of bone tissue resorption after tooth extraction results in significant by changing the initial dimension of the alveolar ridge, due to horizontal and vertical resorption of bone tissue.this process is monitored and by a significant reduction in the volume of soft tissue and the width of the keratinized gingiva.Successful implant therapy is considered when the initial stability is achived of the embedded implant, which largely depends on the width alveolar ridge, at the place of its installation. However, despite achieving the initial stability, inadequate width of the alveolar ridge, and what according to the surgical protocol is a minimum of 1.5 mm. it is the cause of later complications due to present bone resorption processes and peri-implant soft tissue reduction. Regenerative therapy of the horizontal dimension of the alveolar ridge simultaneously with the installation of implants is carried out using biocompatible materials; a basket of thin ones substitutes and collagen membranes. Clinical trials have shown high degree of success of the regenerative therapy of the thinned buccal bone lamella, its deficiencies, as well as occurrences of dehiscence and fenestration, the treatment of which is carried out simultaneously with by inserting an implant. Moreover, simultaneous regenerative therapy of the mentioned bone defects with the installation of implants reduces the risk of buccal bony lamella and soft tissue collapse. Recent review paper and meta-analysis showed complete bony healing of fenestrations and dehiscence regardless of whether a bone substitute with or without collagen is used membrane, which is not the case if the operative region is covered only by mucoperiosteal flap, without regenerative therapy.

The primary goal of this research would be to determine the success of regenerative therapy bone and soft tissue from the buccal side.

ELIGIBILITY:
Inclusion Criteria:

* ASA I classification of health status,

  * Non-smokers or consumption of up to 10 cigarettes per day,
  * No signs of gingival inflammation,
  * Late installation of implants,
  * The possibility of achieving the primary stability of the implant,
  * The dimension of the residual alveolar ridge for implant placement ≥5 mm wide, height ≥12 mm,
  * Diagnosed fenestration, dehiscence of buccal bony lamella ≤3 mm in size and/or thickness of buccal bone lamella ≤1.5 mm,
  * Plaque index (PI) and gingival bleeding on provocation (KNP) <15% and probing depth (DS) <3 mm,
  * Preserved cemento-enamel border (CGG) without the presence of non-carious cervical lesions (NCL), or the presence of a defect in the root area up to 1mm deep with preserved CGG,
  * Preserved interjaw relationships.

Exclusion Criteria:

* Systemic acute administration of drugs up to 7 days before surgical intervention,

  * Systemic chronic administration of steroids or non-steroidal anti-inflammatory drugs,
  * History of oral surgical interventions in the last 4 months,
  * Poor oral hygiene,
  * Demonstrated hypersensitivity to collagen,
  * Pregnancy and breastfeeding,
  * Patient withdrawal from the research protocol in any evaluation period,
  * Patients who underwent standard augmentation of bone tissue with a substitute for bone and membrane, after implant installation,
  * Participation in clinical research in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Achived volume of the bone after implant placement and augmentation | 4 years
  Assessment and comparative analysis quantity of newly formed bone and soft tissue using CBCT and digital, software analysis

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sental Medicine, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Undecided